CLINICAL TRIAL: NCT05204446
Title: Testing a Behavioral Intervention in Pediatric Celiac Disease
Brief Title: Behavioral Intervention for Celiac Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Shayna Coburn, Dr. Shayna Coburn, PhD. Assistant Professor and Attending Psychologist Division of Gastroenterology, Children's National Hospital, George Washington School of Medicine and Health Sciences, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00015490
Record Dates: First submitted 2021-06-14; First posted 2022-01-24 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROW Project (Experimental): ("GROW" Group): Live interactive telehealth-based group meetings will be held for 60 minutes per week over six weeks using Zoom for Telehealth, a HIPAA-compliant platform provided by the PI's institution. A teen group (n=8 per cohort) and a parent group (n=8 per cohort) will be run concurrently but separately, with coordinating topics. Each group meeting will introduce and facilitate discussion of information and CBT-oriented topics for coping and management of CD. Participants will be encouraged to use their audio and video to engage with the interventionist and each other. Between sessions, resources sent through text-based SMS messages using Twilio HIPAA-compliant software 3x/week as reminders of skills and goals for the week.
  Interventions: Behavioral: GROW Project
- Care-As-Usual (No Intervention): Participants assigned to the control group (n=32 dyads) will receive care as usual, which consists of appointments in the Celiac Disease Clinic (at diagnosis, 3 months post-diagnosis, 6 months post-diagnosis, and annually after diagnosis thereafter). These appointments consist of a gastrointestinal physician or nurse practitioner, dietitian, GFD educator, and psychologist for 40-minute consultations each.
- GROW+ Project (Experimental): ("GROW+" Group): Will include the GROW Project with enhanced behavioral strategies and materials identified from phase 2 data (e.g., group discussion about GIP testing, text-based check-ins, etc.) In addition, teens in GROW+ will be encouraged to complete a minimum of 2 GlutenDetect tests per week (12 total) and report results in REDCap (Research Electronic Data Capture, a secure, web-based survey application) throughout the intervention.
  Interventions: Behavioral: GROW+ Project

INTERVENTIONS:
Behavioral: GROW Project — ("GROW" Group): Live interactive telehealth-based group meetings will be held for 60 minutes per week over six weeks using Zoom for Telehealth, a HIPAA-compliant platform provided by the PI's institution. A teen group (n=8 per cohort) and a parent group (n=8 per cohort) will be run concurrently but separately, with coordinating topics. Each group meeting will introduce and facilitate discussion of information and CBT-oriented topics for coping and management of CD. Participants will be encouraged to use their audio and video to engage with the interventionist and each other. Between sessions, resources sent through text-based SMS messages using Twilio HIPAA-compliant software 3x/week as reminders of skills and goals for the week.
  Arms: GROW Project
Behavioral: GROW+ Project — ("GROW+" Group): Will include the GROW Project with enhanced behavioral strategies and materials identified from phase 2 data (e.g., group discussion about GIP testing, text-based check-ins, etc.) In addition, teens in GROW+ will be encouraged to complete a minimum of 2 GlutenDetect tests per week (12 total) and report results in REDCap (Research Electronic Data Capture, a secure, web-based survey application) throughout the intervention.
  Arms: GROW+ Project

SUMMARY:
Celiac disease (CD) is a chronic autoimmune condition whose only currently available treatment is a strict, burdensome gluten-free diet (GFD). The current proposal uses a theory-driven empirical approach for optimizing the GFD for teens and their parents by targeting knowledge, behavior, and coping skills through educational and cognitive-behavioral techniques. Integration with telehealth and SMS (short message service; "text") technology for delivering the intervention has the potential to reduce barriers to specialized treatment at both early and later stages of implementation. The proposed research will refine and test a behavioral intervention for teens with CD and their parents using an iterative stakeholder-centered design. It will consist of a small pilot randomized control trial (RCT) (n=96 dyads) that will examine the preliminary efficacy of the intervention and its impact on quality of life and GFD management by targeting self-efficacy, illness identity, and food-related activities. This work has the potential to make a lasting impact on the standards of care and available treatments to optimize CD management in youth and their families.

DETAILED DESCRIPTION:
Celiac Disease (CD) is an increasingly common disease with significant morbidities if treatment is not achieved. The incidence and prevalence of CD has been increasing in children and teens over the past 15 years in the United States, with prevalence rates nearly tripling from approximately one in 133 to one in fifty children, according to regional population cohort studies. Untreated CD is associated with risks for non-Hodgkin's lymphoma, intestinal cancers, inflammatory bowel disease, diabetes mellitus, and a twofold increase in risks for mortality. The only treatment for CD is a strict Gluten-Free Diet (GFD), which is complex, expensive, tiring, and anxiety-provoking. CD is also associated with impaired quality of life (QOL) and burdensome treatment. Impaired QOL, including poor psychological well-being and functioning, occurs more frequently in CD compared with the general population, likely due to physiological vulnerabilities associated with CD as well as the social impact of the GFD. Teens with CD may experience psychosocial difficulties associated with the GFD due to negative perceptions about reasons for requesting gluten-free foods. Therefore, despite advances in palatable gluten-free products and their availability, youth with CD continue to struggle with GFD management and face new sources of misinformation and misperceptions by others. Like their children, parents are also at risk for poorer QOL resulting from the challenges associated with the treatment of CD in their children. Parents may experience social isolation and stress associated with caring for a child with CD, which can impact family dynamics and the daily tasks of following the GFD. Caregivers who assume responsibility for their children's care report increased depressive symptoms, family stress, and higher burden. According to Social Cognitive Theory, effective support from parents is crucial for successfully managing childhood chronic illnesses and in facilitating the transition to adult medical care, including GFD management. A review of adherence interventions for youth with CD concluded that there is a significant need for evidence-based interventions to support GFD management, and that potential targets should incorporate considerations of the individual, family, community, and health system. The authors also emphasized the promise of novel technologies as a potentially useful and accessible approach for intervention delivery. GIP testing is a promising technology for detecting gluten ingestion, but clinical recommendations and support for GIP testing are needed. GIP testing has demonstrated reliable and valid detection of gluten in relation to histological lesions found via duodenal biopsy as well as high acceptability and feasibility in children and adults. Given the public availability and potential future affordability of GIP test kits, insight into the effects of their use on clinically relevant outcomes is crucial. Additionally, enthusiasm about the potential for accurate biometric assessment of adherence in outcomes research must also be tempered with the possibility that GIP testing may modify behavior and other patient-reported outcomes, with potential benefits or iatrogenic effects. Accordingly, there is an unmet need to counsel patients, particularly teens, on strategies for proactively using at-home GIP tests and optimize outcomes such as QOL and GFD self-management.

The Current Study

The current study is a randomized controlled trial. Participants will total 96 teens (ages 12 to 16 with celiac disease (CD) and their parents or legal guardians (referred to as "parents") who receive medical care from our celiac disease clinics in the Division of Gastroenterology Children's National Hospital (CNH). Dr. Coburn is an integrated member of the Celiac Disease Program Clinical Team, and has met with colleagues, including the gastroenterologist (Dr. Kerzner, Scientific Advisor), nurse, and dietitian, to discuss the proposed study and all team members have expressed their support for this proposal.

After parent-teen dyads have met inclusion criteria, given consent and assent for the RCT, and completed their baseline assessments, the participants will be randomized as dyads into either the "GROW" intervention group, the enhanced "GROW+" intervention group, or the control group. Assignments will be made using block randomization, stratified by the 4 intervention cohorts of 8 dyads each. N=96 parent-teen dyads will be recruited (RCT; 32 in the "GROW" intervention group, 32 in the enhanced "GROW+" intervention group, and 32 in the care-as-usual control group) over the course of the study continuously in cohorts with active recruitment in the investigators' Celiac Disease Clinic as well as through the existing patient database.

Considering the significant challenges faced by teens with celiac disease and their families, there is an urgent need to develop tailored, innovative interventions that are appealing to this age group and potentially efficacious in improving celiac disease-related physiologic and psychosocial functioning. The minimal risks of completing data collection and a 6-week behavioral intervention are reasonable to justify the proposed study, which will minimally provide knowledge on behavioral intervention techniques for teens with CD and their parents and could also lead to improved scientific clarity on the mechanisms that underlie management of special diets in youth. In addition, collection of the psychosocial and clinical data may provide information for health professionals to promote optimal clinical care in youth with celiac disease, with the ultimate goal of reducing risk for long term negative health outcomes. The proposed study has the potential to ultimately result in the availability and implementation of an efficacious intervention for a large community of youth with CD and their families throughout the United States and may have utility in other chronic illness populations as well.

ELIGIBILITY:
Inclusion Criteria:

1. Teens with a physician- confirmed CD diagnosis and one parent or guardian.
2. Teens 12-16 years at the time of enrollment.
3. Proficient in written and spoken English.
4. Have regular access to a device enabled for video conferencing (Zoom) and receiving SMS messages.

Exclusion Criteria:

1. The teen's CD diagnosis is questioned or revoked at any time during the study period;
2. Another member of their household is already enrolled in the study;
3. The teen has a developmental disability or major neuropsychological condition that, in the opinion of the investigators, would impair communication and engagement with the other participants and intervention material.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Teen quality of life as measured by Teen and parent-proxy report on PROMIS Pediatric Profile-37 | Baseline, Immediately Post-Intervention, 3 Month Follow-Up
  Anxiety, depressive symptoms, fatigue, pain interference, physical function-mobility, peer relationships, & pain intensity
Parent quality of life as measured by Parent PROMIS Adult Profile-43 | Baseline, Immediately Post-Intervention, 3 Month Follow-Up
  Parent anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item
Parent health-related quality of life as measured by Parent report PedsQL 2.0 Family Impact Module | Baseline, Immediately Post-Intervention, 3 Month Follow-Up
  Parent impact of child health on quality of life
Teen celiac disease health-related quality of life as measured by Teen self-report on Celiac Disease Quality of Life (CDLIFE) | Baseline, Immediately Post-Intervention, 3 Month Follow-Up
  A validated measure of health-related quality of life in children ages 8-18 living with celiac disease in the United States. 22 items rated 1 (never) to 5 (almost always) for a total possible score ranging from 0-88, with a higher score indicating better health-related quality of life.
Gluten-Free Diet Management (expert) as measured by Expert GFD Adherence Rating (SDE) | Baseline, Immediately Post-Intervention, 3 Month Follow-Up
  Structured global rating by gluten-free diet expert based on dietary recall for potential sources of gluten using online GlutenFreeDiet program.
Gluten-free diet management as measured by Teen & Parent-report Celiac Dietary Adherence Test | Baseline, Immediately Post-Intervention, 3 Month Follow-Up
  Survey measure on symptoms and behavior associated with gluten-free diet management
Gluten Immunogenic Peptides as measured by GlutenDetect | Baseline, Weekly Intervention, Immediately Post-Intervention, 3 Month Follow-Up
  At-home Gluten Detective kit to detect gluten ingested within 24 hours in teen's urine or stool. Teens will be prompted via SMS text message and will be given a 24-hour window to complete the test and send a photo of the results.
Gluten-Free Diet Experiences as assessed by qualitative interview about perceived QOL and GFD management experiences | Baseline, Immediately Post-Intervention, 3 Month Follow-Up
  Semi-structured qualitative interview about current experiences with GFD management for teen/parent.

SECONDARY OUTCOMES:
Self-Efficacy as measured by the Celiac-SE | Baseline, Immediately Post-Intervention, 3 Month Follow-Up
  25-item validated measure of self-efficacy to adhere to the gluten-free diet. Scores below 7 are considered low self-efficacy and scores below 5 indicate very low self-efficacy expectations.
Illness Identity as measured by the Illness Identity Questionnaire | Baseline, Immediately Post-Intervention, 3 Month Follow-Up
  Four illness identity components: rejection, engulfment, acceptance, and enrichment. Agreement rated on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No